CLINICAL TRIAL: NCT03752580
Title: An Investigation to Test a Prototype Nasal Mask in the Home Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-240
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-07

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): Experimental: User Instructions of a Novel Nasal Mask Participants to interpret user instructions in a one hour daytime visit.
  Interventions: Device: User Instructions of novel nasal mask

INTERVENTIONS:
Device: User Instructions of novel nasal mask — User Unstructions interpretation of novel nasal mask for the treatment of obstructive sleep apnea (OSA).

SUMMARY:
This investigation is a prospective non-blinded and non-randomized clinical investigation. This investigation is to test the interpretation of user instructions of a prototype nasal mask on participants. The clinical investigation will be conducted in New Zealand and participants will interact with the user instructions in a one hour daytime visit. A minimum of 15 participants will participate in this trial.

DETAILED DESCRIPTION:
This investigation is to test the interpretation of user instructions of a prototype nasal mask on participants. The clinical investigation will be conducted in New Zealand and participants will interact with the user instructions in a one hour daytime visit. This investigation is designed to evaluate the interpretation by participants of the user instructions. A total number of 20 participants, diagnosed with OSA will be recruited for the trial. The participants will be recruited from the Fisher and Paykel Healthcare Database of subjects (Ethics reference 18/NTA/62).

Fisher and Paykel Healthcare will act as the investigator and sponsor for this investigation. This study will be conducted in accordance with ICH/GCP Guidelines. No deviation from protocol will be implemented without prior review and approval of the sponsor except where it may be necessary to eliminate an immediate hazard to a research participant. In such case, the deviation will be reported to the sponsor (Bhavi Ogra) as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* OSA Mask Users
* 18+ years of age
* Ability to give informed consent

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Mask User Instructions Interpretation | 3 days
  Determined as interpreted by participants from open-ended questions (Open ended questionnaire, very easy - very difficult)- Subjective

CONTACTS AND LOCATIONS:
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand